CLINICAL TRIAL: NCT01025167
Title: The Effect of a New Specific Enteral Formula Compared to a Standard Formula on the Tolerability of a Combined Radio- and Chemotherapy in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Dr. Steffen Benzing, Kabi Innovation Centre, Fresenius Kabi Deutschland GmbH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N-SUP-09-DE
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2010-08

CONDITIONS: Enteral Nutrition
Keywords: cancer; enteral nutrition; omega-3-fatty acids
MeSH Terms: conditions — Neoplasms | interventions — Food

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Test (Experimental): Supportan(R) (500 ml)/disease-specific enteral tube feed for oncologic patients with special key substrates
  Interventions: Dietary Supplement: Supportan(R) (Disease-specific enteral tube feed, food for special medical purposes)
- Control (Placebo Comparator): Fresubin(R) energy fibre (500 ml)/a nutritionally complete enteral standard feed (isoenergetic)
  Interventions: Dietary Supplement: Fresubin(R)

INTERVENTIONS:
Dietary Supplement: Supportan(R) (Disease-specific enteral tube feed, food for special medical purposes) — 500 ml per day / treatment period 11-14 weeks
  Arms: Test
Dietary Supplement: Fresubin(R) — 500 ml/a nutritionally complete enteral standard feed (isoenergetic)
  Arms: Control

SUMMARY:
The purpose of the study is to determine the impact of a specific nutrition formula with a high content of eicosapentaenoic acid (EPA) and fat in oncology patients receiving radio-/chemotherapy on body weight, body composition, nutritional status and physical function compared to a standard nutrition formula. Using an adaptive design approximately 80 patients will be randomized in the first part of the study. Following an interim analysis further 160 patients may be added, for a total of 240 patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with head & neck cancer or oesophagus cancer,
* enteral nutrition with PEG at least for 14 weeks,
* cancer patients who receive a combined radio-/chemotherapy,
* start of nutritional therapy latest at beginning of the radio-/chemotherapy, body mass index >=16 and <=30 kg/m2,0
* Kondrup Score>=3 or SGA = B/C,
* life expectancy > 6 months,
* written informed consent.

Exclusion Criteria:

* second active carcinoma,
* severe diarrhea unresponsive to codeine/loperamide,
* positive anti-HIV-test (safety reasons),
* pregnant or lactating women,
* insulin-dependent diabetes mellitus type I and II,
* patients with cardiac pacemaker,
* allergy to contents of the investigational product, to milk protein or to fish oil,
* patient has no PEG,
* participation in concurrent clinical studies with any other investigational nutritional therapy within one months prior to start of the study,
* intake of muscle growth supportan substances (e.g. anabolics),
* additional fish oil or EPA substitution within the last 4 weeks, SGA status A (well nourished).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2006-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Body cell mass measured by bioelectrical impedance spectroscopy (BIS) | Baseline, mid of radio-/chemotherapy, end of radio-/chemotherapy, day 28 of convalescence period, day 49 of convalescence period

SECONDARY OUTCOMES:
Other parameters of body composition such as fat free mass, lipid mass, total body water, intracellular water, lean tissue mass | Baseline, mid of radio-/chemotherapy, end of radio-/chemotherapy, day 28 of convalescence period, day 49 of convalescence period
Hand grip strength | Baseline, mid of radio-/chemotherapy, end of radio-/chemotherapy, day 28 of convalescence period, day 49 of convalescence period
Quality of Life | Baseline, end of radio-/chemotherapy, day 49 of convalescence period
Gastrointestinal tolerance | Baseline, mid of radio-/chemotherapy, end of radio-/chemotherapy, day 28 of convalescence period, day 49 of convalescence period, daily

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Fietkau, Prof. Dr., Principal Investigator — Department of Radiotherapy University hospital of Erlangen
Locations (10):
- Germany (10):
  - Zentrum für Strahlentherapie und Radioonkologie, Ärztehaus am DIAKO, Bremen
  - Klinik und Poliklinik für Strahlentherapie und Radioonkologie, Universitätsklinikum Dresden, Dresden
  - Department of Radiotherapy, University hospital, Erlangen
  - Klinik für Strahlentherapie und Radioonkologie, Universitätsklinikum Frankfurt, Frankfurt
  - Abteilung Strahlentherapie und Radioonkologie, Universitätsmedizin Göttingen, Göttingen
  - Klinik für Strahlentherapie, Universitätsklinikum Halle, Halle
  - Klinik für Strahlentherapie und Radioonkologie, Universitätsklinikum des Saarlandes, Homburg (Saar)
  - Klinik und Poliklinik für Strahlentherapie Universität Rostock, Rostock
  - Abteilung Strahlentherapie und Radioonkologie, Universitätsmedizin Tübingen, Tübingen
  - Klinik für Strahlentherapie und Radioonkologie, Universitätsklinikum Ulm, Ulm

REFERENCES:
- [Derived] Fietkau R, Lewitzki V, Kuhnt T, Holscher T, Hess CF, Berger B, Wiegel T, Rodel C, Niewald M, Hermann RM, Lubgan D. A disease-specific enteral nutrition formula improves nutritional status and functional performance in patients with head and neck and esophageal cancer undergoing chemoradiotherapy: results of a randomized, controlled, multicenter trial. Cancer. 2013 Sep 15;119(18):3343-53. doi: 10.1002/cncr.28197. Epub 2013 Jun 13. PMID 23765693